CLINICAL TRIAL: NCT01219387
Title: Evaluation of Serum Anti-Mullerian Hormone (AMH) and Inhibin B Levels as Early Predictors of a Successful IVF Cycle in Women Over 38 Years Old.
Brief Title: Evaluation of Anti-mullerian Hormone Levels as Predictive of IVF Outcomes in Women Over 38 Years Old
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Collaborators: Organon (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RMA-00-09
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: AMH Levels; Inhibin B Levels; IVF Patients Over 38 Years Old
Keywords: AMH; inhibin B; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The present study is designed to evaluate the basal serum levels of anti-mullerian hormone (AMH) and inhibin B as early predictors of ovarian response, implantation rate, and pregnancy rate in women 38 years old or older that are undergoing an IVF cycle.

DETAILED DESCRIPTION:
Specifics aims are: a) to describe AMH and inhibin levels on day 3 previous to ART cycle; b) to analyze the association between these hormone levels and the retrieved metaphase II oocytes quantity; c) to analyze the association between these hormone levels and quality embryo score d) to analyze the association between these hormone levels and the number of gestational sacs per transferred-embryo (implantation rate); e) to analyze the association between these hormone levels and the pregnancy rate; f) to make a prediction model for pregnancy rate by using a multivariable regression analysis.

Patient participation includes signing the consent and having additional tubes of blood drawn at a regularly scheduled blood draw. This blood is used to run the study tests (AMH and inhibin levels).

ELIGIBILITY:
Inclusion Criteria:

1. Women 38 years old or older at the time of initiating treatment

Exclusion Criteria:

1. Uterine disease: malformation, septum, submucosal myomas, endometrial polyps Advanced endometriosis with endometrioma (s)
2. No uterus
3. Single ovary

Ages: 38 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing IVF treatment who are over the age of 38 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
AMH levels as predictive of oocyte quality | within 3 months
  Evaluate the relationship between a patients AMH and inhibin level prior to beginning IVF treatment and the oocyte quality as observed during the IVF cycle
AMH levels as predictive of embryo quality | within 3 months
  Evaluate the relationship between a patients AMH and inhibin level prior to beginning IVF treatment and the embryo quality as observed during the IVF cycle
AMH levels as predictive of implantation and pregnancy outcomes | 1 year
  Evaluate the relationship between a patients AMH and inhibin level prior to beginning IVF treatment and rates of implantation and delivery during that IVF cycle

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Bergh, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (2):
- United States (2):
  - Reproductive Medicine Assoicates of New Jersey, Morristown, New Jersey
  - Reproductive Medicine Associates of PA at Lehigh Valley, Allentown, Pennsylvania